CLINICAL TRIAL: NCT05359874
Title: Improvement of the Operative Outcome in Patients With Primary VEGF Positive Unifocal Breast Cancer or Ductal Carcinoma in Situ (DCIS) Through the Intraoperative Visualization of the Tumor Using Molecular Imaging and Fluorescent Markers Bevacizumab-IRDye-800CW
Brief Title: Improvement of the Operative Outcome in Patients With Primary VEGF + Unifocal Breast Cancer or DCIS Through the Intraoperative Visualization of the Tumor Using Molecular Imaging and Bevacizumab-IRDye-800CW
Acronym: DoT-FMI
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: application has been withdrawn
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOT-1871-KIE-0120-I
Record Dates: First submitted 2021-05-14; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental)
  Interventions: Drug: Bevacizumab-IRDye800CW

INTERVENTIONS:
Drug: Bevacizumab-IRDye800CW — In order to be able to detect this marker in vivo, special multispectral fluorescence-reflecting cameras (MFRI) were developed, which can be used for the intraoperative display of the tumor and potentially affected lymph nodes and which are now to be evaluated together with the fluorescence marker.
  Other Names: Device: special multispectral fluorescence-reflecting cameras

SUMMARY:
It is a prospective, open, non-randomized, multicenter, one-armed, blinded (surgeon), diagnostic clinical trial according to AMG and MPG. The fluorescent marker Bevacizumab-IRDye800CW has advantages over conventional methods of tumor imaging in terms of accuracy, patient safety and validity. In order to be able to detect this marker in vivo, special multispectral fluorescence-reflecting cameras (MFRI) were developed, which can be used for the intraoperative display of the tumor and potentially affected lymph nodes and which are now to be evaluated together with the fluorescence marker.

DETAILED DESCRIPTION:
Complete surgical excision of the tumor (R0 resection) is the cornerstone of any curative therapy concept for cancer. In order to be able to achieve the highest possible rate of R0 resections, the tumor, its localization and spread needs to be more precisely represented. This should be possible through an intraoperative representation of the tumor by means of fluorescence imaging at the molecular level.

Vascular Endothelial Growth Factor (VEGF, or VEGF-A), which is expressed differently in normal and tumor tissue, is a suitable marker for molecular imaging, especially in gynecological cancer. Bevacizumab is a genetically engineered humanized monoclonal antibody that is directed against VEGF and is already therapeutically approved for the treatment of breast and ovarian cancer and has also shown efficacy in studies on endometrial cancer.

Fluorescence-labeled bevacizumab has advantages over conventional methods of tumor imaging in terms of accuracy, patient safety, cost efficiency and validity. A fluorescent marker, Bevacizumab-IRDye800CW, was developed and recently used in clinical trials in the Netherlands. In order to be able to detect this marker in vivo, special multispectral fluorescence-reflecting cameras (MFRI) were developed, which can be used for intraoperative visualization of the tumor and potentially affected lymph nodes. These systems can now be used to evaluate the fluorescent marker in clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* women of age ≥ 18 years able to give consent who have been informed in detail about the study beforehand and have given written consent to participate
* Patients with histologically confirmed unifocal VEGF-positive invasive breast cancer with an indication for BET
* Patients with histologically confirmed unilateral VEGF-positive DCIS with an indication for BET
* ECOG performance ≤ 2
* Pre-menopausal women had a negative pregnancy test prior to administration of the study medication
* Negative pregnancy test (serum) within 10 days prior to administration of the test medication in all women of childbearing age with results available prior to the start of therapy (or postmenopausal; age ≥60 and no menses over ≥ 1 year without any other medical cause; or hysterectomy, or tube ligation, or bilaterally guided occlusion). Women of childbearing potential who are sexually active must agree that they and their partner may use effective contraception during the trial and for 3 months after participation

Exclusion Criteria:

* Second malignancy in the breast and other organs
* Pregnant or breastfeeding patients
* Planned sentinel lymph node marking using patent blue
* Previous radiation therapy in the area to be examined
* Known or suspected hypersensitivity to the study medication (according to IMPD / SmPC) or other immunoglobulins
* Currently after neoadjuvant (primarily systemic) chemotherapy and anti-hormone therapy
* Immunotherapy (e.g. monoclonal antibodies, cytokines or signal transduction inhibitors) in the last 28 days prior to the declaration of consent
* Previous therapy with bevacizumab
* Planned reconstruction in the breast to be examined
* Previous surgery within the last 28 days prior to the declaration of consent
* Non-healing wounds, ulcers or broken bones within the last 28 days prior to giving informed consent
* Patients with ileus within the last 28 days prior to the declaration of consent
* Non-adjustable hypertension (> 145/90 mmHg) despite optimal drug therapy
* Insufficient kidney function (serum creatinine> 1.5 x upper limit of the normal range)
* Current or recent treatment with another investigational drug in another clinical trial within 28 days of informed consent
* Potentially fertile women without adequate contraception. Safe contraceptive measures are procedures with a Pearl index of ≤ 1%
* Patients with other serious illnesses that pose an unreasonable risk for participating in the study
* Persons who are in a dependent / employment relationship with the sponsor or investigator
* Persons who are to be or are to be accommodated in an institution due to a court or official order

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Determination of the sensitivity and specificity of bevacizumab- IRDye800CW | 21 days
  Determination of the sensitivity and specificity of bevacizumab- IRDye800CW with regard to the identification of the tumor margins compared with the histopathological findings (resection result R0, R1) as the gold standard

SECONDARY OUTCOMES:
Safety and Toxicity of Bevacizumab-IRDye800CW will be analyzed by absolute and relative frequencies of Safety events | 21 days
  Absolute and relative frequencies of AE, SAE, AR, and SAR are presented by MedDRA System Organ Class and Preferred Term.

IPD SHARING:
Plan to Share IPD: Undecided
no patient specific data will be shared